CLINICAL TRIAL: NCT07161765
Title: Rectal Evacuation Disorders and Straining-associated Symptoms in Bleeding Hemorrhoids
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Shah, Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00275895; R03DK143921-01 (NIH)
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Bleeding Hemorrhoids; Rectal Evacuation Disorders
Keywords: Anorectal testing; Rectal Expulsion Device (RED)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Rectal Expulsion Device (Experimental)
  Interventions: Device: Rectal Expulsion Device (RED)

INTERVENTIONS:
Device: Rectal Expulsion Device (RED) — Enrolled participants will complete surveys prior a standard of care visit at the University of Michigan.
  Gastroenterology staff will perform the RED device at the time of a participant's anorectal manometry appointment.

SUMMARY:
This study aims to understand the mechanisms of straining on anorectal testing, to better help people receive more effective treatment advice. The study also aims to understand how point-of-care anorectal testing with an FDA-cleared device called Rectal Expulsion Device (RED) helps to identify people that might benefit from specific treatments that target pelvic floor muscle problems that lead to straining and hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

* Participants had a colonoscopy within the last 12 months for rectal bleeding (with no cause of bleeding found other than hemorrhoids).
* Participants provider placed an order for anorectal manometry to the University of Michigan

Exclusion Criteria:

* Anal fissure
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Intra-class correlation (ICC) between overall Patient Assessment of Constipation Symptom Score (PAC-SYM) and Hemorrhoid Disease Symptom Score (HDSS) sum scores | Day 1 (standard of care clinic visit)
  The PAC-SYM survey has 12 questions in which participants select from Absent (0)-Very severe (4) There is a range of scores from 0-48 with a higher score indicating more severe symptoms.
  The HDSS survey has 5 questions in which participants select from Never (0)- Every day (always) (4).
  There is a range of scores from 0-20 with a higher score indicating more severe symptoms.
  ICC will be assessed between overall PAC-SYM and Hemorrhoid Disease Symptom Score (HDSS) sum scores, with a value of >0.70 considered acceptable. A sample size of 100 patients is typical to achieve a minimum acceptable ICC of 0.70 with a confidence interval of 0.10.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Shah, MD, Principal Investigator — University of Michigan
Locations (1):
- University of MIchigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No